CLINICAL TRIAL: NCT07087054
Title: A Randomized, Parallel Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Paltusotine in Adults With Carcinoid Syndrome Due to Well-Differentiated Neuroendocrine Tumors
Brief Title: Carcinoid Syndrome Efficacy Study Featuring an Oral Daily Paltusotine Regimen
Acronym: CAREFNDR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRN00808-12; 2024-519875-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-09; First posted 2025-07-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Carcinoid Syndrome; Carcinoid; Carcinoid Tumor; Carcinoid Tumor of Ileum; Carcinoid Tumor of Cecum; Carcinoid Tumor of Liver; Carcinoid Tumor of Pancreas; Carcinoid Syndrome Diarrhea; Carcinoid Intestine Tumor
Keywords: Neuroendocrine tumor; Paltusotine; CRN00808; Carcinoid syndrome; Lanreotide; Octreotide; Somatostatin agonist
MeSH Terms: conditions — Serotonin Syndrome; Carcinoid Tumor; Carcinoid Tumors, Intestinal; Neuroendocrine Tumors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paltusotine 80 mg daily (Experimental)
  Interventions: Drug: Paltusotine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paltusotine — Experimental Drug: Randomized
  Arms: Paltusotine 80 mg daily
Drug: Placebo — Matching Placebo Drug: Randomized
  Arms: Placebo

SUMMARY:
A Phase 3, randomized, double-blinded, placebo-controlled study to evaluate the efficacy and safety of paltusotine treatment vs placebo as well as the long-term safety of paltusotine in adults with carcinoid syndrome due to well-differentiated neuroendocrine tumors. The purpose of this study is to continue the evaluation of the safety, efficacy, and pharmacokinetics (PK) of paltusotine in participants with carcinoid syndrome.

DETAILED DESCRIPTION:
This is a global, randomized, parallel-group, placebo-controlled study to evaluate the efficacy and safety of paltusotine in adults with carcinoid syndrome. The study includes a screening period of up to 11 weeks, a double-blinded randomized control period of 16 weeks, an open label extension period of 104 weeks, and a follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age, at the time of Screening.
* Willing and able to comply with the study procedures as specified in the protocol, including at least 70% compliance with the study diary for the 2-week period.
* Documented carcinoid syndrome requiring medical therapy. Participants must exhibit symptoms of flushing with or without frequent BMs as follows:

  * For participants who are naïve/not currently treated with somatostatin receptors ligands (SRL), they must exhibit an average of >1 flushing episode/day over a period of 14 days
  * For participants who will wash out from SRL treatment, they must exhibit an increase in daily average flushing episodes and an average of >1 flushing episode/day over a period of 14 days during the Washout Period.
* Evaluable documentation of locally advanced or metastatic histopathologically confirmed well-differentiated neuroendocrine tumor(s) [NETs].
* No significant disease progression as assessed by the Investigator within the last 6 months before randomization.

Exclusion Criteria:

* Diarrhea attributed to any condition(s) other than carcinoid syndrome.
* Uncontrolled/severe diarrhea associated with significant volume contraction, dehydration, or hypotension.
* Requires second line treatments (eg, telotristat) for control of carcinoid syndrome symptoms in the opinion of the Investigator.
* Treatment with specific NET therapy <4 weeks before Screening (such as everolimus or sunitinib) or hepatic embolization, radiotherapy, peptide receptor radionuclide therapy (PRRT), and/or tumor debulking <12 weeks before Screening.
* Major surgery within 8 weeks before Screening.
* History of another primary malignancy <3 years prior to the date of randomization, except for adequately treated basal or squamous cell carcinoma of the skin, cancer of the breast or cervix in situ, previously treated malignancy, if all treatment for that malignancy was completed at least 3 years prior to first dose of study treatment, and no current evidence of disease, concurrent malignancy determined to be clinically stable and not requiring treatment.
* Diabetes mellitus treated with insulin for less than 6 weeks prior to the study entry.
* Poorly controlled diabetes mellitus defined as having a hemoglobin A1c (HbA1c) ≥8.5%
* Unable to administer short-acting (SA) octreotide (octreotide acetate injection), or prior nonresponse documented with somatostatin agonists.
* Clinically significant concomitant disease or indicator of disease that is not a result of the primary disease under study, including but not limited to cardiovascular disease, estimated glomerular filtration rate 2×upper limit of normal [ULN], and/or total bilirubin (TB) >1.5×ULN. (Participants with previously diagnosed Gilbert's syndrome not accompanied by other hepatobiliary disorders and associated with TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Participants will record the number of flushing per day in a daily diary to assess the efficacy of paltusotine vs placebo in reducing flushing episodes. | Measured at Week 12
  Treatment group difference of change from baseline to Week 12 in flushing episodes/day averaged over the 14 days prior to Week 12.

SECONDARY OUTCOMES:
Participants will record the number of bowel movements (BMs) per day in a daily diary to assess the efficacy of paltusotine vs placebo in reducing BMs/day. | Measured at Week 12
  Treatment group difference of change from baseline to Week 12 in BMs/day averaged over the 14 days prior to Week 12.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (10):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Yale University - New Haven Hospital - Yale Cancer Center, New Haven, Connecticut
  - Winshop Cancer Institute - Emory University, Atlanta, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Louisiana State University Health Sciences, Metairie, Louisiana
  - Henry Ford Cancer - Detroit, Detroit, Michigan
  - Mayo Clinic, Rochester, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
- Argentina (4):
  - Sanatorio Guemes, Buenos Aires
  - Centro de Endocrinologia y Diabetes Dr. A. Gutman ICM - Investigaciones, Buenos Aires
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires
  - Instituto Médico de la Fundación Estudios Clínicos, Santa Fe
- Brazil (3):
  - AC Camargo Cancer Center, São Paulo, Brazil
  - Sociedade Literaria e Caritativa Santos Agostinho - Hospital Sao José, Criciúma
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
- France (6):
  - CHRU Tours - Hopital Trousseau, Chambray-lès-Tours
  - Hopital Beaujun - APHP, Clichy
  - APHM- Hopital de la Timone, Marseille
  - Centre Hospitalier Universitaire Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Bordeaux - Hopital Haut-Leveque, Pessac
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No